CLINICAL TRIAL: NCT03831802
Title: Quality of Life in Epilepsy Patients Wearing a Biosensor for Seizure Detection Through Electrodermal Activity and Accelerometry - a Pilot Study
Brief Title: Embrace and Quality of Life
Acronym: EMBQL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because of technical issues
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Philippe Ryvlin, Head of Department of Clinical Neurosciences, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMBQL
Record Dates: First submitted 2018-08-21; First posted 2019-02-06 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Epilepsy, Tonic-Clonic
Keywords: epilepsy; mhealth; quality of life
MeSH Terms: conditions — Epilepsy, Tonic-Clonic; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): The experimental group will make use of the Alert app that sends alarms to patients mobile devices, and if desired to the mobile devices of their caregivers. This group will also use the Mate app which is used as a seizure diary
  Interventions: Device: Embrace with Alert and Mate apps
- Control group (Active Comparator): The control group will only use the Mate app and not the Alert app. This group will thus not receive any notification, from the device, and will be unaware, of the devices performance
  Interventions: Device: Embrace with Mate app only

INTERVENTIONS:
Device: Embrace with Alert and Mate apps — Patients will wear the device on their wrist as often as possible during the day and night. The Embrace Watch contains sensors and memory recordings of electrodermal activity, temperature and physical activity from the wearer. This group will receive notifications on the mobile phone when seizure takes place. Quality of life questionnaires will be filled by the patients at the first follow-up and final assessments.
  Other Names: experimental group's intervention
  Arms: experimental group
Device: Embrace with Mate app only — Patients will wear the device on their wrist as often as possible during the day and night. This group will just use the Mate app that summarizes Embrace Watch data for the owner and captures contextual information around events.This group will not receive any alert notification on the mobile phone when a seizure takes place.
  Other Names: Control group's intervention
  Arms: Control group

SUMMARY:
A prospective, open, randomized, pilot clinical trial which aims the assessment of quality of life (QOL) in epilepsy outpatients equipped with a wrist-worn biosensor that provides measures of electrodermal activity and accelerometry. These measures are used to automatically detect epileptic seizures that are transmitted to a mobile phone-based system for alerts and recording.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged >18 years old
* clearcut diagnosis of epilepsy without evidence of non epileptic psychogenic seizure
* primary tonic clonic seizures or focal seizures evolving to generalized tonic clonic convulsion
* seizure frequency > 1 seizure/month during the last three months
* signed the informed consent form
* own a mobile phone device compatible with the embrace apps
* able to use the device without help from caregivers

Exclusion Criteria:

* patients aged less than 18 years old
* epilepsy diagnosis remains uncertain
* evidence of psychogenic non epileptic seizures
* seizure frequency below 1/month during any of the three previous months
* past-history of nickel allergy and contact dermatitis
* did not sign the informed consent form
* does not own mobile phone device compatible with the embrace apps
* cognitive or behavioral impairment preventing compliance or correct use of the device and app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
The mean change from Baseline of the total score, of the french version of the Quality of life Epilepsy inventory-31 | 3 month
  The change between the QOLIE-31 questionnaire total score measured at the first and the final visit will serve as primary endpoint. The possible range of each scale's final score is from 0 to 100. higher scores reflect better quality of life.

SECONDARY OUTCOMES:
The mean change from Baseline of the total scores of seven Quality of Life in Epilepsy Inventory-31 subscales covering the following epilepsy-specific domains: | 3 month
  Epilepsy-specific domains are: seizure worry, overall QOL, emotional well being, energy/fatigue subscales, medication effects, work-driving-social limits, cognitive function subscales. The possible range of each scale's final score is from 0 to 100. Higher scores reflect better quality of life.
Total number of true and false positives seizure detection | 3 month
  Detected by the embrace device, saved via the alert app and controlled by the patient via the mate app
The usability total score of Embrace and Mate apps | 3 month
  Will be assessed with the System usability scale (SUS). The score are to 0 from 100.
The utility total score of the system in general | 3 month
  will be assessed via a structured questionnaire-based interview that was Tailored for this study

CONTACTS AND LOCATIONS:
Locations (1):
- Neurotech, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No